CLINICAL TRIAL: NCT05078892
Title: Fertility Attitudes of Adolescents and Young Adults With Turner Syndrome and Their Parents/Guardians (The Fertility ConcepTS Study)
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000335; 000335-CH
Record Dates: First submitted 2021-10-14; First posted 2021-10-15 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Fertility Perservation; Fertility
Keywords: Phenotyping; attitudes of individuals with TS; survey of adolescents and young adults; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adolescents (12-17): Adolescents 12-17 with Turner Syndrome
- Parents of Adolescents (12-17): Parents of Adolescents (12-17)with Turner Syndrome
- Young Adults (18-25): Young Adults (18-25)with Turner Syndrome

SUMMARY:
Background:

Turner syndrome (TS) is caused by the partial or complete absence of one of the two X

chromosomes in all cells or a portion of cells. Adolescents and young adults (AYAs) with TS and their families are not routinely counseled about fertility issues and options. Researchers want to learn more about the attitudes of AYAs with TS and their parents or guardians regarding future fertility.

Objective:

To create and distribute a survey for AYAs with TS and their parents or guardians that will improve understanding about their attitudes toward fertility, fertility preservation, and options for building a family.

Eligibility:

Female AYAs aged 12-25 years with TS, and parents or guardians of AYAs with TS.

Design:

Participants will be put into 3 focus groups: females ages 12-17 with TS; females ages 18-25 with TS; and parents or guardians of AYAs with TS. Each focus group session will be held via Zoom. Participants can use video or just audio for the session. They will use their first name. If they prefer, they can use a pseudonym. Each group will meet once. The session will last 90 minutes.

Participants will receive a draft of the survey. The survey questions ask about fertility and pregnancy. Participants will evaluate the usefulness and relevance of each question. They will be asked if any question should be changed. The survey will be finalized based on their feedback. The final survey will be distributed through TS groups.

Participation will last for 1 day....

DETAILED DESCRIPTION:
This study aims to improve our understanding of attitudes of adolescents and young adults (AYA) with Turner Syndrome and their parents/guardians towards fertility, fertility preservation, and options for building a family through development and dissemination of a fertility attitudes questionnaire.

Primary Objective: To compare differences in attitudes between AYA with TS and their parents regarding survey content area (i) medical/surgical fertility preservation procedures with unknown outcomes.

Secondary Objectives:

1. To compare differences in attitudes between AYA with TS and their parents regarding survey content areas (ii) interest in understanding the effects of TS on fertility and pregnancy and (iii) opinions of having children that are genetically similar and alternative methods of building a family.
2. To compare differences in attitudes between adolescents aged 12-17 years and young adults aged 18-25 years with TS regarding survey content areas (i) medical/surgical fertility preservation procedures with unknown outcomes, (ii) interest in understanding the effects of TS on fertility and pregnancy, and (iii) opinions of having children that are genetically similar and alternative methods of building a family.

Primary Endpoint: Difference in response scores between AYA with TS-parent dyads to the survey questions addressing survey content area (i) interest in medical/surgical fertility preservation procedures with unknown outcomes.

Secondary Endpoints:

1. Differences in response scores between AYA with TS-parent dyads to the survey questions addressing survey content areas

   (ii) interest in understanding the effects of TS on fertility and pregnancy, and (iii) opinions of having children that are genetically similar and alternative methods of building a family.
2. Differences in response scores between adolescents with TS ages 12 to 17 years and young adults with TS ages 18 to 25 years to the survey content areas addressing (i) interest in medical/surgical fertility preservation procedures with unknown outcomes, (ii) interest in understanding the effects of TS on fertility and pregnancy, and (iii) opinions of having children that are genetically similar and alternative methods of building a family

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration ofthe study
2. Adolescents and young adults ages 12 to 25 years who self- identify as having Turnersyndrome
3. Individuals who self-identity as parents/guardians of adolescents and young adults ages12 to 25 years with Turner syndrome

EXCLUSION CRITERIA:

Inability to read and comprehend written and Verbal English as the surveys required for the study have not been translated for non-English speaking subjects.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: For the three focus groups, participants will consist of adolescents and young adults with Turner Syndrome and their parents/guardians recruited from members of the Turner Syndrome Global Alliance (TSGA) by their leadership. An IRB-approved flyer will be sent to the TSGA for distribution to their members. The Fertility Attitudes survey will be disseminated by various TS support groups through a link for the survey webpage and an IRB-approved flyer with a QR code and link to an online survey webpage via the Clinical Trials Survey System (CTSS) provided to their members via their email as well as through their social media site (Facebook page).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
SURVEY CONTENT | Baseline
  To compare differences in survey response scores between adolescents/young adults with TS and their parents regarding survey content areas (i) medical/surgical fertility preservation procedures with unknown outcomes.
SURVEY CONTENT | Baseline
  Differences in attitudes between AYA with TS and their parents regarding survey content area (i) medical/surgical fertility preservation procedures with unknown outcomes

SECONDARY OUTCOMES:
RESPONSE SCORES | Baseline
  Differences in responses between AYA with TS and their parents to the survey content
RESPONSE SCORES | Baseline
  Differences in responses between adolescents aged 12-17 years and young adults aged 18-25 years with TS regarding survey content

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Gomez-Lobo, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institute of Child Health and Human Development (NICHD), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
.The protocol does not have a plan for IPD at this time.